CLINICAL TRIAL: NCT01897792
Title: Effect of Antioxidant Vitamins on Coagulopathy and Nosocomial Pneumonia After Severe Trauma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit patients that meet inclusion criteria.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jean-Francois Pittet, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F101108001
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Coagulopathy; Nosocomial Pneumonia
MeSH Terms: conditions — Hemostatic Disorders; Healthcare-Associated Pneumonia | interventions — Ascorbic Acid; Vitamin E; alpha-Tocopherol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamins C and E (Experimental): Vitamin C (1,000 mg i.v.) and Vitamin E (1,000 IU p.o. via the naso-gastric tube) administered every 8 hours starting within one hour after admission to the Emergency department for up to 5 days or until discharge from the ICU, whichever comes first.
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin E
- 0.9% saline and sugar pill (Placebo Comparator): 100 ml of 0.9% saline (for i.v. Vitamin C) and a p.o. placebo (sugar pill for the p.o. Vitamin E) administered every 8 hours starting within one hour after admission to the Emergency department for up to 5 days or until discharge from the ICU, whichever comes first.
  Interventions: Dietary Supplement: Saline (for Vitamin C); Drug: Placebo (for Vitamin E)

INTERVENTIONS:
Dietary Supplement: Vitamin C
  Other Names: ascorbic acid
  Arms: Vitamins C and E
Dietary Supplement: Vitamin E
  Other Names: alpha-tocopherol
  Arms: Vitamins C and E
Dietary Supplement: Saline (for Vitamin C) — 0.9% saline administered to mimic Vitamin C
  Arms: 0.9% saline and sugar pill
Drug: Placebo (for Vitamin E) — Sugar pill administered to mimic Vitamin E
  Arms: 0.9% saline and sugar pill

SUMMARY:
The purpose of this study is to determine the effect of antioxidant vitamins (vitamins C and E) on the development of coagulation derangements and nosocomial pneumonia after severe trauma in patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients admitted to the emergency department at the University of Alabama at Birmingham (UAB) Hospital
* Blunt or penetrating injury
* UAB highest trauma activation

Exclusion Criteria:

* Age < 19 years of age
* Patients with known bleeding diathesis or who are concurrently taking anticoagulant medication
* Patients with known liver disease
* Minor patients
* Pregnant patients (known or suspected pregnancy)
* Patients who are incarcerated
* Patients who lack a surrogate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Pittet, M.D., Principal Investigator — The University of Alabama at Birmingham; Jeffrey Kerby, M.D., Ph.D., Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham Hospital, Birmingham, Alabama, United States

REFERENCES:
- [Background] Brohi K, Cohen MJ, Ganter MT, Matthay MA, Mackersie RC, Pittet JF. Acute traumatic coagulopathy: initiated by hypoperfusion: modulated through the protein C pathway? Ann Surg. 2007 May;245(5):812-8. doi: 10.1097/01.sla.0000256862.79374.31. PMID 17457176
- [Background] Brohi K, Cohen MJ, Ganter MT, Schultz MJ, Levi M, Mackersie RC, Pittet JF. Acute coagulopathy of trauma: hypoperfusion induces systemic anticoagulation and hyperfibrinolysis. J Trauma. 2008 May;64(5):1211-7; discussion 1217. doi: 10.1097/TA.0b013e318169cd3c. PMID 18469643
- [Background] Chesebro BB, Rahn P, Carles M, Esmon CT, Xu J, Brohi K, Frith D, Pittet JF, Cohen MJ. Increase in activated protein C mediates acute traumatic coagulopathy in mice. Shock. 2009 Dec;32(6):659-65. doi: 10.1097/SHK.0b013e3181a5a632. PMID 19333141
- [Background] Cohen MJ, Bir N, Rahn P, Dotson R, Brohi K, Chesebro BB, Mackersie R, Carles M, Wiener-Kronish J, Pittet JF. Protein C depletion early after trauma increases the risk of ventilator-associated pneumonia. J Trauma. 2009 Dec;67(6):1176-81. doi: 10.1097/TA.0b013e3181c1c1bc. PMID 20009664
- [Background] Nathens AB, Neff MJ, Jurkovich GJ, Klotz P, Farver K, Ruzinski JT, Radella F, Garcia I, Maier RV. Randomized, prospective trial of antioxidant supplementation in critically ill surgical patients. Ann Surg. 2002 Dec;236(6):814-22. doi: 10.1097/00000658-200212000-00014. PMID 12454520
- [Background] Collier BR, Giladi A, Dossett LA, Dyer L, Fleming SB, Cotton BA. Impact of high-dose antioxidants on outcomes in acutely injured patients. JPEN J Parenter Enteral Nutr. 2008 Jul-Aug;32(4):384-8. doi: 10.1177/0148607108319808. PMID 18596309
- [Background] Secor D, Li F, Ellis CG, Sharpe MD, Gross PL, Wilson JX, Tyml K. Impaired microvascular perfusion in sepsis requires activated coagulation and P-selectin-mediated platelet adhesion in capillaries. Intensive Care Med. 2010 Nov;36(11):1928-34. doi: 10.1007/s00134-010-1969-3. Epub 2010 Aug 6. PMID 20689935
- [Background] Brohi K, Singh J, Heron M, Coats T. Acute traumatic coagulopathy. J Trauma. 2003 Jun;54(6):1127-30. doi: 10.1097/01.TA.0000069184.82147.06. PMID 12813333
- [Background] MacLeod JB, Lynn M, McKenney MG, Cohn SM, Murtha M. Early coagulopathy predicts mortality in trauma. J Trauma. 2003 Jul;55(1):39-44. doi: 10.1097/01.TA.0000075338.21177.EF. PMID 12855879
- [Background] Esmon CT. The protein C pathway. Chest. 2003 Sep;124(3 Suppl):26S-32S. doi: 10.1378/chest.124.3_suppl.26s. PMID 12970121
- [Background] Giladi AM, Dossett LA, Fleming SB, Abumrad NN, Cotton BA. High-dose antioxidant administration is associated with a reduction in post-injury complications in critically ill trauma patients. Injury. 2011 Jan;42(1):78-82. doi: 10.1016/j.injury.2010.01.104. Epub 2010 Feb 10. PMID 20149369

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamins C and E: Vitamin C (1,000 mg i.v.) and Vitamin E (1,000 IU p.o. via the naso-gastric tube) administered every 8 hours starting within one hour after admission to the Emergency department for up to 5 days or until discharge from the ICU, whichever comes first.
  Vitamin C
  Vitamin E
Period: Overall Study
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Coagulation Abnormalities
Description: Coagulation parameters are evaluated using standard functional tests (prothrombin time (PT), partial thromboplastin time (PTT), fibrinogen and platelet count)and point of care functional analysis using thromboelastogram (TEG-ROTEM). A blood sample is collected upon arrival in the emergency department at 0 hours only and analyzed for markers of activation of coagulation, inflammation, and levels of vitamin C/E.
Time Frame: From enrollment up to 3 days
Measure: Number; unit: participants
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
participants | 2 | 1

2. Primary Outcome: Number of Subjects With Ventilator-associated Pneumonia.
Description: Number of subjects diagnosed with pneumonia and requiring ventilator support.
Time Frame: From enrollment to 3 days
Measure: Number; unit: participants
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
participants | 4 | 2

3. Primary Outcome: Number of Subjects With Organ Injury
Description: Any injury to internal organs (thoracic, abdominal or cranial cavity)
Time Frame: From enrollment to 3 days
Measure: Number; unit: participants
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
participants | 0 | 0

4. Primary Outcome: Number of Total Blood Product Transfusions
Description: the number of blood product transfusions for all subjects in each group over the course of 3 days.
Time Frame: From enrollment to 3 days
Measure: Number; unit: blood transfusions
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
blood transfusions | 11 | 5

5. Secondary Outcome: Number of Protocol Violations Per Arm.
Description: The number of times that there was a deviation or violation from how the protocol was to be implemented.
Time Frame: from enrollment up to 60 days post enrollment
Measure: Number; unit: protocol deviations
Groups:
- Vitamin C and E Participants -; 0.9% Saline and Sugar Pill Participants - Protocol Violations: # of protocol deviations
Arm/Group | Vitamin C and E Participants - | 0.9% Saline and Sugar Pill Participants - Protocol Violations
Number analyzed (Participants) | 6 | 5
protocol deviations | 1 | 0

6. Secondary Outcome: Number of Subjects Surviving to Day 28
Description: Number of subjects that survived to day 28 after enrollment
Time Frame: from enrollment up to 28 days post enrollment
Measure: Number; unit: participants
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
participants | 6 | 5

7. Secondary Outcome: Number of Subjects With 60-day Survival
Description: Number of subjects in each arm that survived to day 60
Time Frame: from enrollment up to 60 days post enrollment
Measure: Number; unit: participants
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
participants | 6 | 5

8. Secondary Outcome: Mean Number of Ventilator-free Days for Subjects
Description: The mean number of ventilator free days (not on ventilator) for subjects in each arm
Time Frame: from enrollment up to 60 days post enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
days | 12 [2 to 23] | 6.2 [1 to 17]

9. Secondary Outcome: Mean Number of Days in ICU.
Description: the mean number of days each subject was in the ICU in each arm
Time Frame: from enrollment up to 60 days post enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
days | 15 [3 to 30] | 11 [4 to 20]

10. Secondary Outcome: Mean Number of Hospital Stay Days.
Description: The mean number of days subjects were in the hospital in each arm of the study
Time Frame: from enrollment up to 60 days post enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Number analyzed (Participants) | 6 | 5
days | 18.3 [6 to 39] | 18.2 [6 to 26]

ADVERSE EVENTS:
Description: No adverse events were collected
Arm/Group | Vitamins C and E | 0.9% Saline and Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated--inability to recruit patient that met inclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes